CLINICAL TRIAL: NCT06830434
Title: Aesthetic Crown Lengthening: Laser Impact on Pain Perception and Surgery Impact on Self-esteem and Quality of Life Perceptions
Brief Title: Aesthetic Crown Lengthening: Laser Impact on Pain Perception and Perceptions on Self-esteem and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22735519.9.0000.5418
Record Dates: First submitted 2020-10-05; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2020-10

CONDITIONS: Crown Lengthening; Pain Postoperative; Self Concept
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Twenty patients will be selected based on their interest in undergoing aesthetic crown lengthening surgery in the anterior maxillary region and their indication for the procedure. Two questionnaires will be administered: the OHIP-14/Brazil and the Rosenberg Self-Esteem Scale - UNIFESP/EPM. In one study arm, laser therapy will be performed in a blinded manner immediately after the surgical procedure.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Laser therapy will be performed in a blinded manner for the patients. The crown lengthening surgeon and the outcomes assessor will also be blinded-they will not know which side received the laser therapy. Only the laser operator will have access to this information. The quadrant receiving the therapy will be randomly selected using a computer program by the laser operator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crown lenghtening surgery associated with Laser therapy (Experimental): After crown lenghtening surgery in aesthetic area, the laser will be applied on the "Right" or "Left" oral side (chosen randomly), in all the 20 patients, in a "Split-mouth" model.
  Interventions: Procedure: Crown lengthening surgery
- Crown lenghtening surgery without Laser therapy (Placebo Comparator): After crown lenghtening surgery in aesthetic area, all the 20 patients, will not receive laser treatment on an oral side.
  Interventions: Procedure: Crown lengthening surgery

INTERVENTIONS:
Procedure: Crown lengthening surgery — Following clinical and radiographic examinations and thorough case planning, surgical procedures were performed under local anesthesia by a single operator. After anesthesia, the distance from the gingival margin to the cementoenamel junction will be measured, and these values will be transferred to the gingival tissue to guide the procedure. Excess gingival tissue will be excised, and, when necessary, an osteotomy will be performed to re-establish the supracrestal attachment tissues.

SUMMARY:
Gummy smile is a condition that promotes a disharmonious smile, altering confidence and decreasing self-esteem of many patients. Luckily, this problem in most cases is easily solved by aesthetic crown lengthening surgery. However, this is a surgery that is still considered by many patients to be painful and uncomfortable. Thereby, this study seeks both to evaluate possible changes in patients' self-esteem and self-confidence after the aesthetic crown lengthening surgery.

DETAILED DESCRIPTION:
Periodontally healthy patients who expressed interest in undergoing ACL will be selected. Before surgery, two questionnaires will be administered: the OHIP-14/Brazil and the Rosenberg Self-Esteem Scale-UNIFESP/EPM. These tools are designed to assess patients' perceptions of self-esteem and quality of life and will be re-administered 30 days and one year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Periodontal health diagnosis (full mouth bleeding on probing - BP <10%, clinical attachment level - CAL ≤ 3mm),
* Distance from the gingival margin to the cementum-enamel junction ≥ 3mm associated with a gingival smile and / or short clinical crowns when compared to anatomical crowns, due to the altered passive eruption or gingival overgrowth).
* Good general health

Exclusion Criteria:

* Presence of systemic changes (diabetes, heart disease, hepatitis, etc.)
* Use of medications (such as antibiotics, continuous anti-inflammatory drugs, phenytoin, cyclosporine) that may influence the response to the surgical treatment
* Diagnosis of gingivitis and/or periodontitis
* Smoking habit
* Pregnancy or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Patients' levels of self-esteem and quality of life | From enrollment through study completion, an average of 2 years
  The perceptions of self-esteem and quality will be measured through the OHIP-14/Brazil and the Rosenberg/UNIFESP-EPM Self-Esteem Scale questionnaires.The Rosenberg questionnaire addresses an individual's overall sense of self-worth and self-acceptance, evaluating both positive and negative self-perception domains to provide a holistic view of their self-esteem. It consists of 10 statements rated on a 4-point Likert scale, with responses ranging from 'Strongly Agree' to 'Strongly Disagree.' Scores range from 0 to 30, where higher scores indicate greater self-esteem, while lower scores suggest diminished self-worth or a negative self-view. The OHIP-14 (Oral Health Impact Profile-14) questionnaire evaluates the impact of oral health on an individual's quality of life. It measures functional and psychological well-being across seven domains to assess how oral conditions affect daily life and overall well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campinas, UNICAMP, Piracicaba, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No